CLINICAL TRIAL: NCT06517160
Title: A Randomised Controlled Trial to Compare MedBook Portal and Standard Care in Medication Reconciliation at Transitions of Care From Hospital Discharge to Primary Healthcare Settings
Brief Title: Comparison of MedBook Portal and Usual Care in Medication Reconciliation at Primary Healthcare Upon Hospital Discharge
Acronym: MEDRECON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Phang Yen Yen, Principal Investigator/ Senior Principal Assistant Director (Pharmacy Practice & Development), Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRR-22-02409-ODX
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Medication Reconciliation
Keywords: Medication Reconciliation; Medication Safety; Unintentional Medication Discrepancies; Primary Healthcare; Transition of Care; Electronic Health Record

STUDY DESIGN:
Masking Description: Doctors at health clinics were not aware of the subjects in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients will receive standard care, where doctors review previous medical records in the home-based medical card and discharge notes if provided by the patient during their first review. Doctors cannot access the patient's discharge medication list from the MedBook Portal, and no MedBook Portal Notice is attached to the patient's home-based medical card.
  The principal investigator will give a list of control group patients to the study pharmacist at the health clinic. Knowing their appointment dates, the study pharmacist will search for the first prescription after transitioning care from the hospital to the primary health clinic. The study pharmacist will then compare the discharge prescription in the MedBook Portal with the first prescription to identify medication discrepancies. Any discrepancies will be addressed by confirming with the doctor whether they are intentional or unintentional.
- Intervention Group (Experimental): MedBook Portal Notice will be attached to the patient's home-based medical card for doctors and pharmacists at health clinics to identify recruited patients during their first follow-up after hospital discharge. During the doctor's review of intervention group patients, the doctor will log in to the MedBook Portal to check the discharge medication list and review the case based on the previous medical record in the home-based medical card and the discharge note, if provided. The doctor will then conduct medication reconciliation by comparing the discharge prescription with the new prescription. Study pharmacists at health clinics will screen patients' home-based medical cards when collecting medications. Study pharmacists will retrieve the discharge prescription from the MedBook Portal and conduct medication reconciliation by comparing the discharge prescription with the new prescription. Any discrepancies will be addressed by confirming with the doctor whether they are intentional.
  Interventions: Other: MedBook Portal

INTERVENTIONS:
Other: MedBook Portal — Intervention Group (With MedBook Portal & MedBook Portal Notice)
  1. MedBook Portal Notice in front of the patient home-based medical card
  2. Discharge prescriptions are uploaded into MedBook Portal and can be retrieved by doctors & pharmacists.
  MedBook portal (https://aplikasi.jknsarawak.moh.gov.my/medbook) is a webpage that enable sharing of patient medication records among healthcare facilities under Ministry of Health. Sarawak State Health Department owned and managed this portal. All the information is kept under their server. Doctors in the Health Clinics and Study Pharmacists will be given access to this portal whereby each of the healthcare providers shall log in using their Identification Number and the password created by them. Doctor shall log in to MedBook Portal to check on discharge medication list when reviewing the patient at health clinic. MedBook Portal can be accessed both using a smartphone or a computer.
  Arms: Intervention Group

SUMMARY:
A randomized controlled trial was conducted to examine the efficacy of the MedBook portal in reducing medication discrepancies after discharge. The MedBook portal is a webpage that enables the sharing of patient medication profiles among healthcare facilities under the Ministry of Health. A total of 398 adult patients in general medical wards, who were discharged from Sarawak General Hospital, Sibu Hospital, Miri Hospital, and Sarikei Hospital, and referred to ten public primary health clinics located near these hospitals, were recruited for this study. Eligible subjects were randomized into an intervention group and a control group in a 1:1 ratio. This study was conducted from May 2023 to July 2024.

Study pharmacists conducted medication reconciliation before randomization by comparing the discharge prescription with the pre-admission medications and inpatient medication charts to identify discrepancies. Discrepancies were confirmed with the doctor to determine if they were intentional or unintentional.

Control group patients received standard care, with discharge notes and appointment dates provided upon discharge. In Malaysia, there is no shared electronic medication record system between primary and secondary healthcare; thus, information is transferred manually via discharge notes and home-based medical cards. During initial health clinic visits, doctors reviewed patients' medical records based on home-based medical cards and discharge notes, if available. Pharmacists conducted medication reconciliation by comparing new prescriptions with previous records. Discrepancies were confirmed with the doctor to determine if they were intentional or unintentional. Control group doctors could not access the MedBook Portal, and no MedBook Portal Notice was attached to home-based medical cards.

The MedBook Portal Notice was attached to patients' home-based medical cards for identification at follow-up appointments. Doctors logged into the MedBook Portal to access discharge medication lists and conducted medication reconciliation by comparing discharge prescriptions with new prescriptions. Study pharmacists screened patients' home-based medical cards at the pharmacy, identified recruited patients via the MedBook Portal Notice, and conducted medication reconciliation by comparing new prescriptions with discharge medication lists in the portal. Discrepancies were confirmed with the doctor to determine if they were intentional or unintentional.

DETAILED DESCRIPTION:
Study Design, Population and Setting This prospective, multicentre randomised controlled trial compared the prevalence of medication discrepancies in the first prescription upon transition of care from hospitals to primary health clinics between MedBook Portal and standard care. The MedBook portal is a webpage that enables the sharing of patient medication records among healthcare facilities under Ministry of Health. Doctors in the health clinics and pharmacists log in to MedBook Portal to check the discharge medication list when reviewing the patient at the clinic. The study adhered to the Consolidated Standards of Reporting Trials (CONSORT) Statement guideline, employing a 1:1 allocation ratio allocation ratio to two groups: the intervention group and the control group.

The targeted population was the adult patients in Sarawak who were discharged from the public tertiary or secondary hospitals, including Sarawak General Hospital, Sibu Hospital, Sarikei Hospital, and Miri Hospital, and referred to ten public primary health clinics located nearby these hospitals. The ten public primary health clinics were Batu Kawa Health Clinic, Kota Sentosa Health Clinic, Kota Samarahan Health Clinic, Jalan Oya Health Clinic, Lanang Health Clinic, Sibu Jaya Health Clinic, Miri Health Clinic, Tudan Health Clinic, Sarikei Health Clinic, and Bintangor Health Clinic.

Data collection took place over a year from May 2023 to July 2024. The research was granted with ethical approval by the Medical Research &amp; Ethics Committee (MREC), Ministry of Health Malaysia [NMRR-22-02409-ODX (IIR)].

This study enrolled adult patients aged 18 years and older who were admitted to general medical wards who had comorbidities related to cardiovascular, renal, respiratory, or endocrine system, as well as patients referred to the selected primary health clinics after hospital discharge and possessed home-based medical cards. Patients discharged during public holidays or weekends were excluded.

Medication Reconciliation Upon Hospital Discharge The discharge prescription served as the primary reference for discharge reconciliation, as it contained the list of medications that the pharmacy would use for preparation and dispensing to patients upon discharge. Study pharmacists conducted discharge medication reconciliation before randomisation. This process involved comparing the medications listed in the discharge prescription with those documented in the medication history assessment form (representing pre-admission medications) and the inpatient medication charts (representing medications initiated during admission) to identify any discrepancies before preparing the discharge medications. If any disparities were found, study pharmacists confirmed with the doctor to determine whether they were intentional or unintentional medication discrepancies, with any amendments documented on the discharge prescription.

Randomisation and blinding The recruited patients were randomised into the intervention and control groups in a 1: 1 ratio before discharge. Randomisation was conducted using an online program available at http://www.graphpad.com/quickcalcs/index.cfm. A research coordinator was appointed to administer the randomisation and inform the study pharmacist to deliver the intervention according to the assigned group. The research coordinator had no direct contact with patients, study pharmacists and doctors. Additionally, the research coordinator managed the patient list, including their assigned codes and group allocation. Subsequently, the research coordinator sent the patient list to the principal investigator to remind the patient of the follow-up dates at the health clinic. Due to the nature of the intervention, neither patients, doctors, nor study pharmacists were blinded to the group assignments.

Control Group The control group received standard care, where upon discharge, patients were provided with discharge notes by nurses along with their appointment dates at the health clinics. In Malaysia, there is currently no shared electronic medication record system between primary and secondary healthcare; hence, information on medical history and medication history has to be transferred manually via discharge note and home-based medical card. During their initial visit at the health clinic, doctors reviewed patients' medical records based on information from their home-based medical cards and discharge notes, if provided by the patient. Pharmacists at the health clinics conducted medication reconciliation by comparing the new prescriptions received against the patients' previous medical records in their home-based medical cards and discharge notes, if available. Any identified discrepancies were addressed through confirmation with the doctor to determine whether they were intentional or unintentional.

In contrast, doctors in the control group were unable to access a patients' discharge medication list from the MedBook Portal, and no MedBook Portal Notice was attached to the patients' home-based medical card. The principal investigator provided a patient list in the control group to the study pharmacist at the health clinic. By knowing their appointment date, the study pharmacist searched for the first prescription upon transitioning care from the hospital to the primary health clinic. Subsequently, the study pharmacist compared the discharge prescription in MedBook Portal with the first prescription to identify any medication discrepancies. If discrepancies were found, study pharmacists confirmed with the doctor to determine whether they were intentional or unintentional. However, the study pharmacist might not be able to retrieve the first prescription immediately on the appointment date due to the absence of a MedBook Portal Notice. Consequently, the study pharmacist could only address any identified discrepancies with the prescriber at a later time.

Intervention Group The MedBook Portal Notice was attached to the patient's home-based medical card to enable doctors and pharmacists at health clinics to identify the recruited patients. This appointment would be their first follow-up at health clinics after discharge from the hospital.

During the doctor's review of the patient in the intervention group, the doctor logged into the MedBook Portal to access the discharge medication list and reviewed the case based on the previous medical record in the home-based medical card and the discharge note, if provided by the patient during their first visit. Subsequently, the doctor conducted medication reconciliation by comparing the list of medications in the discharge prescription against the new prescription prepared.

At the health clinics, study pharmacists screened patients' home-based medical cards presented at the pharmacy when collecting medications. Upon identifying the recruited patients via the MedBook Portal Notice, pharmacists logged into the MedBook Portal to access the discharge medication list. They then conducted medication reconciliation by comparing the new prescription received against the discharge medication list in the portal. Interventions were carried out by the study pharmacists through confirmation with the doctor to determine whether any identified medication discrepancies were intentional or unintentional.

Operational Definitions Medication discrepancy is defined as any variation or difference in medication regimen identified when comparing an old medication list with newly prescribed medications. Intentional medication discrepancy is a justified discrepancy due to a change in the patient's clinical condition. Unintentional medication discrepancy is an unjustified discrepancy identified after checking with prescriber and it is a medication error, specifically prescribing error Medication discrepancies are classified discrepant dose, discrepant frequency, polypharmacy, drug omission, drug addition, and inappropriate drug.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and above in general medical wards.
* Patients who had any of the following comorbidities: (1) cardiovascular related diseases, e.g.: hypertension, acute coronary syndrome, heart failure, stroke, atrial fibrillation; (2) endocrine related diseases, e.g.: diabetes, thyroid disorders; (3) renal related diseases, e.g.: chronic kidney disease, end stage renal failure; (4) respiratory related diseases, e.g.: asthma, chronic obstructive pulmonary disease.
* Patients who are referred to the selected primary health clinics after hospital discharge.
* Patients with home-based medical card.

Exclusion Criteria:

• Patients discharged during public holidays or weekends will be excluded from this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Percentage of prescriptions with medication discrepancies in the first prescription during the first follow-up visit at the primary health clinic after hospital discharge | From enrollment to the first appointment date at the selected primary health clinic, the time frame might range from 1 week to 2 months
  (Number of prescription with medication discrepancies during 1st health clinic follow up)/(Total prescription reconcilled at health clinic (with or without MedBook Portal))

SECONDARY OUTCOMES:
Percentage of prescriptions with medication discrepancies in the discharge prescription | From enrollment to hospital discharge, time time frame might range from 1 hour to 2 days.
  Number of prescription with medication errors/ Total prescription reconcilled upon discharge
Type of medication discrepancies | From enrollment to the first appointment date at the selected primary health clinic, the time frame might range from 1 week to 2 months
  Number of medication discrepancies detected will be grouped into 0, 1, 2, 3, 4, 5 errors. Chi-square test will be used to analyse the association of medication discrepancies at intervention group versus control group.
Predictors associated with medication discrepancies | From enrollment to the first appointment date at the selected primary health clinic, the time frame might range from 1 week to 2 months
  Multiple logistic regression

CONTACTS AND LOCATIONS:
Overall Officials: Yen Yen Phang, Principal Investigator — Sarawak State Health Department
Locations (1):
- Sarawak State Health Department, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No
No personal information will be disclosed and subjects will not be identified when the findings of the study are published. However, Study Protocol and Informed Consent Form, data are available upon reasonable request from the corresponding author.

REFERENCES:
- [Derived] Phang YY, Kuan JW, Oh AL, Ting CY, Osman NA, Moses S. Effectiveness of digital platform in reducing unintentional medication discrepancies at transition of care from hospital discharge to primary healthcare settings: a randomised controlled trial. BMC Prim Care. 2025 Jul 2;26(1):206. doi: 10.1186/s12875-025-02904-z. PMID 40604512
- See also: This study was registered with the Medical Research & Ethics Committee, Ministry Of Health Malaysia, under registration number NMRR ID-22-02409-ODX (IIR) on 30 November 2022. — https://nmrr.gov.my/research-directory/0e78f0f4-5b02-411e-bbb5-33d60cb273d0

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT06517160/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT06517160/ICF_002.pdf